CLINICAL TRIAL: NCT04250415
Title: Prospective, Multi-Center Adolescent Clavicle Fracture Registry
Brief Title: Multi-Center Adolescent Clavicle Fracture Trial: Operative vs. Non-Operative Treatment
Acronym: FACTS
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Rady Children's Hospital, San Diego (Other); University of Michigan (Other); Texas Scottish Rite Hospital for Children (Other); Washington University School of Medicine (Other); Campbell Clinic (Other); University of California, San Francisco (Other); Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Benton Heyworth, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00004816
Record Dates: First submitted 2020-01-23; First posted 2020-01-31 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Clavicle Fracture
Keywords: Adolescent
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Operative Arm
  Interventions: Procedure: Surgery
- Non-operative Arm

INTERVENTIONS:
Procedure: Surgery
  Groups: Operative Arm

SUMMARY:
Investigators from eight tertiary care, level 1 pediatric trauma centers have developed a protocol for the establishment of a formal, prospective multi-center adolescent clavicle registry, with designs for standardized radiographic assessment and the prospective collection of validated outcome measures and complications data, for all patients, ages 10-18, treated for clavicle shaft fractures, operatively and non-operatively. Eventually, the investigators would like to do comparative analysis for the operative and non-operative treatment arms, with additional sub-stratified analyses performed within these treatment arms by age and activity level. Among the primary goals of research projects stemming from the first arm of this registry, FACTS A, is to explore the hypothesis that non-operative treatment is associated with lower costs, greater safety, and equivalent or superior outcomes, compared with operative treatment, despite a national trend towards increasing surgical treatment. The second arm of the registry, FACTS B, will continue to investigate the same hypotheses, excluding cost outcomes, in patients only with completely displaced midshaft clavicle fractures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10-18
* Diagnosis of a primary diaphyseal clavicle fracture
* Fracture must be completely displaced
* Patient - BCH subjects must pursue follow-up at BCH main campus or Waltham must be 59 days or less from the primary fracture
* All study patients (across all sites) must agree to be contacted by a long-term follow-up coordinator based out of Boston Children's Hospital for long-term follow-up questions (out to the 2-year time point). This can/will be done via phone, mail, text message, and/or email.

Exclusion Criteria:

* Pathological fracture
* Previous ipsilateral fracture
* Unable to fill out outcome collection forms
* Refusal to participate
* Underlying neurologic or neurocognitive disorder that affects UE function
* Underlying metabolic bone disorder (e.g. osteogenesis imperfecta) that significantly alters normal bone healing
* Unable to project injury X-ray films if treated initially at an institution that is not a member of this register

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Males and females between the ages of 10 and 18, who visit Boston Children's Hospital or one of the other participating institutions for treatment of a primary, completely displaced mid-shaft clavicle fracture.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-03-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in functional score from time of injury (or from time of surgery) using the American Shoulder and Elbow Surgeons score (ASES) | 2 years
  Patient-reported function over time will be assessed using the American Shoulder and Elbow Surgeons score (ASES).
  The ASES is a composite instrument comprised of two sections, including patient self-reported pain (7 items) and patient self-reported activities of daily living (10 items). Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.

SECONDARY OUTCOMES:
Changes in functional score from time of injury (or from time of surgery) using the Disabilities of the Arm, Shoulder, and Hand Score (Quick-DASH). | 2 years
  Patient reported function over time will be assessed using the Disabilities of the Arm, Shoulder, and Hand Score (Quick-DASH).
  The QuickDASH questionnaire evaluates presence and degree of symptoms as well as perceived ability to perform functional tasks with the injured upper extremity. There are 5 responses for each question, graded on a scale from '1' to '5'. A response of '1' reflects the patient's perception to have either 'no symptoms', no limitations, or no perceived disability to the question prompt. A response of '5' reflects the patient's perception to have either 'extreme' symptoms, or inability to perform the task prompted in the question.
Changes in Activity Level from time of injury (or from time of surgery) using the Marx Shoulder Activity Scale. | 2 years
  Patient-reported activity level over time will be assessed using the Marx Shoulder Activity Scale.
  This questionnaire rates the frequency for which a patient is able to perform five functional activities with the injured upper extremity. Each prompt is rated on a five-point frequency scale from 'never performed' (0 points) to 'daily' (4 points). Two additional questions regarding ability to participate in sports generally considered 'contact sports' and ability to participate in sports involving 'overhead throwing' are rated on a scaled from 'No' (0 points) to 'Yes, on a professional level' (3 points). A higher cumulative score is reflective of 'better' function.
Patient Quality of Life after injury (or surgery) using the EQ-5D-3L. | 2 years
  Patient reported quality of life will be assessed through distribution of the EQ-5D-3L questionnaire. The EQ-5D-3L questionnaire is comprised from 5 dimensions including: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Responses are scored on an algorithm in which a higher number is indicative of a greater quality of life.
Patient Quality of Life after injury (or surgery) using the EQ-VAS. | 2 years
  Patient reported quality of life will be assessed through distribution of the EQ-VAS questionnaire. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state' ranging from the numerical value of '100' ('Best imaginable health state') to '0' ('Worst imaginable health state'). The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Patient Satisfaction with treatment outcome after injury (or surgery) | 2 years
  Patients will be asked a series of 'yes-no' questions as well as questions related to their clinical progression since time of treatment for which responses range from 'completely satisfied' to 'completely unsatisfied'. If a patient underwent internal fixation with implanted hardware, the patient will be asked whether or not the hardware is bothersome.
  The rate of choice selection for each response, per question, will be cumulatively assessed.
Patient Return-to-Sport after injury (or surgery) | 2 years
  Patients will be asked their ability to return to sporting activities and level of competition compared to before their clavicle injury. Self-reported athletes will be further queried as to what sport/s they returned to, and whether they returned to the same level of competition. If athletes have not returned to play, or have returned at a less competitive level, they will be asked whether the change in sport participation or sport intensity was related to the clavicle injury, or due to other circumstances.
  The rate of choice selection for each response, per question, will be cumulatively assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Benton E Heyworth, MD, Principal Investigator — Boston Children's Hospital
Locations (8):
- United States (8):
  - University of California San Francisco Benioff Children's Hospital Oakland, Oakland, California
  - Rady Children's Hospital, San Diego, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Washington University at St. Louis, St Louis, Missouri
  - Campbell Clinic Orthopaedics, Memphis, Tennessee
  - Texas Scottish Rite Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heyworth BE, Pennock AT, Li Y, Liotta ES, Dragonetti B, Williams D, Ellis HB, Nepple JJ, Spence D, Willimon SC, Perkins CA, Pandya NK, Kocher MS, Edmonds EW, Wilson PL, Busch MT, Sabatini CS, Farley F, Bae DS. Two-Year Functional Outcomes of Operative vs Nonoperative Treatment of Completely Displaced Midshaft Clavicle Fractures in Adolescents: Results From the Prospective Multicenter FACTS Study Group. Am J Sports Med. 2022 Sep;50(11):3045-3055. doi: 10.1177/03635465221114420. Epub 2022 Aug 19. PMID 35984091